CLINICAL TRIAL: NCT07358897
Title: Gender Affirming Hormone Therapy and Immune Function in Trans Individuals - The GIFT Study
Acronym: GIFT
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 182929; 361618 (Other: Integrated Research Application System)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Transgender

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will keep peripheral blood mononuclear cells, stabilised whole blood and serum and plasma samples for 10 years after the study has completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our immune systems protect us from infection but can also cause disease, for example by attacking our own bodies (autoimmune disease), or driving chronic inflammation in conditions such as heart disease. The immune systems of men and women function differently, as evidenced by differing rates of disease with autoimmune disease being more common in women whilst men are more susceptible to infection. We don't know why these differences exist, but if we could understand we may be able to develop new treatments to treat or prevent immune driven diseases. So far, we know that both sex chromosomes and hormones affect how the immune system functions, but not the exact contribution of each or how they interact. One way to study this is to work with transgender people. Transgender people identify as a gender different from their sex assigned at birth and some may choose to take the sex hormones of the gender they identify with, which is known as gender affirming hormone therapy (GAHT). Given that these changes affect their sex hormone profile and not their chromosomes, any changes in their immune system would be driven by hormones only. This would help us understand not only how sex hormones shape the immune system more generally, but also the disease risk in transgender people and enable better patient counselling. In this study, transgender patients starting on GAHT at 56 Dean Street clinic in London would be invited to donate blood samples before starting therapy, at 1 month (optional) and at 3 and 6 months. These samples would be analysed at the Laboratory of Medical Sciences to examine how the different types of immune cells change with therapy and how they respond to different immune triggers (stimuli). We aim to recruit 500 individuals and anticipate the study will last up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 50 years of age with diagnosed gender dysphoria about to start gender-affirming hormone therapy with either oestrogen or testosterone.

Exclusion Criteria:

* Lack of capacity to consent.
* Abnormalities in expected pubertal development and pharmacological interventions that could affect levels of gonadal steroids including suspected or confirmed self-treatment with steroid hormone preparations in preceding month (birth control excluded).
* Serious immunological disease (immune deficiency, autoimmune disease requiring immunomodulatory treatment).
* Regular immunomodulatory treatment such as prednisolone or biological drugs.
* In the case of vaccination or symptomatic infection ≤5 days before the visit blood sampling should be postponed by 1 week.
* Age <18 years or >50 years
* Completed menopause (persons assigned female sex at birth).
* Positivity for blood borne viruses (HIV, Hepatitis B, Hepatitis C, HTLV-1)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults between 18 and 50 years of age with diagnosed gender dysphoria about to start gender-affirming hormone therapy with either oestrogen or testosterone.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2029-01-07 (Estimated); Study Completion 2029-01-07 (Estimated)

PRIMARY OUTCOMES:
Immune system adaptations to gender affirming hormone therapy | 3 years
  We will measure how immune system populations change quantitatively (i.e. the relative proportions of each subpopulation) and in their responses to different immune stimuli with gender affirming hormone therapy.

SECONDARY OUTCOMES:
Hormone concentrations | 3 years
  We will measure blood sex hormone levels of individuals on gender affirming hormone therapy
Immune-related blood protein levels | 3 years
  We will measure concentration of immune related proteins in plasma samples from patients on gender affirming hormone therapy